CLINICAL TRIAL: NCT03316755
Title: Risk Perception of Periodontal Disease: A Randomised Clinical Trial
Brief Title: Risk Perception of Periodontal Disease
Acronym: RPPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Benin (Other)
Responsible Party: Principal Investigator, Clement Chinedu Azodo, Head of Department, University of Benin
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Perio
Record Dates: First submitted 2017-10-09; First posted 2017-10-20 (Actual); Last update posted 2017-10-20 (Actual); Status verified 2017-10

CONDITIONS: Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Intervention Model Description: randomised
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- without pamphlet (No Intervention): a group not exposed to pamphlet
- With pamphlets (Experimental): a group exposed to pamphlet
  Interventions: Behavioral: Exposure

INTERVENTIONS:
Behavioral: Exposure — Exposure to pamphlet
  Arms: With pamphlets

SUMMARY:
This study aimed at understanding the impact of educational pamphlet on Risk Perception of Periodontal Disease using A Randomised Clinical Trial model among patients in a Nigerian outpatient dental clinic

DETAILED DESCRIPTION:
This study aimed at understanding the impact of educational pamphlet on Risk Perception of Periodontal Disease using A Randomised Clinical Trial model among patients in a Nigerian outpatient dental clinic. The outcome will help activate a success oriented periodontal disease prevention model

ELIGIBILITY:
Inclusion Criteria:

* consenting dental patients

Exclusion Criteria:

* non consenting dental patients

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 300 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-10-04 (Actual); Study Completion 2017-10-07 (Actual)

PRIMARY OUTCOMES:
Risk perception | 1month
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Clement C Azodo, Principal Investigator — UBTH
Locations (1):
- UBenin, Benin City, Edo, Nigeria

IPD SHARING:
Plan to Share IPD: Undecided